CLINICAL TRIAL: NCT02793752
Title: A Prospective Study to Determine if Mitochondrial Activity of Cumulus Cells From the Cumulus-oocyte Complex is Associated With Maternal Age and Oocyte Competence to Blastocyst
Brief Title: Mitochondrial Activity of Cumulus Cells From the Cumulus-oocyte Complex and Oocyte Competence
Status: Completed | Type: Observational
Sponsor: Main Line Fertility Center (Other)
Responsible Party: Sponsor
Other Study IDs: MLFC-005
Record Dates: First submitted 2016-06-03; First posted 2016-06-08 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Infertility
Keywords: IVF; In vitro fertilization; Cumulus Cells; Oocyte; Embryo; Fertility
MeSH Terms: conditions — Infertility | interventions — Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cumulus Cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mitochondrial Activity of Cumulus Cells: One way that cumulus cells influence oocyte competence is via metabolism (Dumesic et al., 2015). Analysis of mitochondria respiration is an established methodology used for evaluation of cell metabolic homeostasis and for diagnosis of different pathologies.
  Interventions: Other: Age
- Competence to Blastocyst: The percentage of fertilized eggs that develop to the blastocyst stage.
  Interventions: Other: Age

INTERVENTIONS:
Other: Age — Maternal Age

SUMMARY:
The need for non-invasive biomarkers of oocyte competency has become urgent as women increasingly delay attempts at childbearing. The aging process is complex and includes impaired mitochondrial dysfunction, oxidative stress, diminished metabolic activity, and activity of several cell-signaling systems. Cumulus cells form an intimate association with the oocyte in the follicle, and they can have a significant impact on oocyte meiotic and developmental competence. In the IVF lab, the clump of cumulus cells is typically cut away from the oocyte immediately after an oocyte retrieval procedure, and then the cumulus cells are discarded. Measuring the mitochondrial respiratory activity of cumulus cells may serve as a non-invasive biomarker for oocyte competency and a predictor of reproductive success in IVF patients in the future.

DETAILED DESCRIPTION:
Background The number of couples undergoing in vitro fertilization (IVF) is rapidly growing worldwide. However, only approximately 5% of aspirated human oocytes have the competence to implant and develop into a child (Ziebe, 2013). Reasons for this low percentage of competence include genetic abnormalities and metabolic problems.

Moreover, this oocyte developmental competence decreases as a woman ages, and therefore maternal age is the single best predictor of reproductive outcome in women (Keefe et al, 2015). In general, the aging process is complex and includes impaired mitochondrial dysfunction, oxidative stress, diminished metabolic activity, and activity of several cell-signaling systems (Bentov, 2011).

Oocyte Competency is the Key to Embryo Potential The oocyte is the major determinant of embryo developmental competence in women. The oocyte transmits not only the mother's nuclear but also her mitochondrial genome to the embryo. The maternal and paternal genomes are neither symmetrical nor equal in their contributions to embryo fate.

Oxygen Consumption and Oocyte/Embryo Competence Clinically useful biomarkers of oocyte competency are needed (Keefe et al, 2015). Oxygen consumption is a quality marker for human oocyte competence conditioned by ovarian stimulation regimens (Tejera et al., 2011). Furthermore, oxygen consumption rates of embryos have been found to be associated with successful implantation and can be used to select the embryo with the best developmental potential (Tejera et al., 2012).

Rationale of Studying Cumulus Cells Ovarian follicles are highly specialized structures that support the growth and development of oocytes during controlled ovarian stimulation for IVF. Cumulus cells are somatic cells that form an intimate association with the oocyte in the follicle. Cumulus cells possess specialized cytoplasmic projections that penetrate through the zona pellucida [shell] and form gap junctions at their tips with the oocyte, generating an elaborate structure called the cumulus-oocyte complex (COC) (Albertini et al., 2001; Gilchrist et al., 2008). Cumulus cells metabolize the bulk of the glucose consumed by the COC to supply metabolic intermediates to the oocyte, and COC glucose metabolism is pivotal in determining oocyte developmental competence (Sutton-McDowall et al., 2010). It is well known that cumulus cells support oocyte development through the provision of essential nutrients, information molecules, metabolic precursors and signaling molecules (Hutt et al., 2007). Because of the metabolic and communication link between the cumulus and the oocyte, glucose availability and metabolism within the cumulus can have a significant impact on oocyte meiotic and developmental competence (Thompson JG, 2007).

If the coordinated somatic cell-oocyte interactions are perturbed by metabolic disease and/or maternal aging, molecular damage of the oocyte can alter macromolecules, induce mitochondrial mutations, all of which can harm the oocyte (Dumesic et al, 2015). For example, in 2015 Hsu et al. reported that endometriosis may be associated with mitochondrial dysfunction in pooled cumulus cells, and subjects with endometriosis may have a defect in cumulus cell mitochondrial function, which may contribute to decreased fertilization and implantation rates (Barnhart et al., 2002). The purpose of this study is to determine if the mitochondrial respiratory activity of cumulus cells is associated with maternal age and reproductive outcomes (oocyte competence).

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing IVF in an attempt to achieve pregnancy.
2. Day 3 FSH < 10 IU/ml, LH< 12 IU/ml, and estradiol <50 pg/ml on day 2-4 of menstrual cycle
3. Antimullerian Hormone > 1.5 and < 10
4. Between 10 and 20 basal antral follicles on day 2-4 of the menstrual cycle
5. Body weight >50 kg, with BMI > 18 and < 32 kg/m2

Exclusion Criteria:

1. Smokers
2. Polycystic ovarian disease
3. Endometriosis greater than Stage I
4. Testicular or Epididymal Sperm
5. PGD/PGS

Ages: 21 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients undergoing in vitro fertilization
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-03; Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Mitochondrial respiration of cumulus Cells | Day of cumulus collection
Blastocyst development | Five to six days after fertilization

CONTACTS AND LOCATIONS:
Overall Officials: Sharon H Anderson, PhD, Study Director — Main Line Fertility Center
Locations (1):
- Main Line Fertility Center, Bryn Mawr, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: website for Main Line Fertility — http://mainlinefertility.com